CLINICAL TRIAL: NCT01240512
Title: Daylight: The Effect of Vitamin D Supplementation on Blood Pressure in Vitamin D Deficient Individuals With Pre-Hypertension
Brief Title: DAYLIGHT: Vitamin D Therapy in Individuals at High Risk of Hypertension
Acronym: DAYLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hartford Hospital (Other); Allina Health System (Other)
Responsible Party: Principal Investigator, Thomas J. Wang, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010P001612
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Vitamin D Deficiency; Pre-Hypertension
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency; Prehypertension | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Arm (Active Comparator): 4000 IU/day Vitamin D3 (cholecalciferol) supplementation
  Interventions: Drug: Cholecalciferol
- Low Dose Arm (Active Comparator): 400 IU/day Vitamin D3 (cholecalciferol) supplementation
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D3 (cholecalciferol) 200 IU and 2000 IU drops will be supplied by D Drops. It is supplied as a liquid containing 400 drops/bottle with a potency of 200 IU/drop or 2000 IU/drop. The contents of the label will be in accordance with all applicable regulatory requirements. The droppers are gravity-metered to deliver a consistent drop size (dosage). Two drops (either 200 IU or 2000 IU) of Vitamin D (cholecalciferol) is to be taken orally once-daily.
  Other Names: Vitamin D3

SUMMARY:
This is a randomized, double-blind, multicenter, 6-month follow-up trial of low (400 IU/day) versus high (4000 IU/day) dose vitamin D supplementation in individuals with pre- and early stage 1 hypertension and vitamin D deficiency. A total of 530 participants (265 participants per treatment arm) will be randomized between 3 sites. Approximately 2,250 participants will be screened between the 3 sites. Vital signs, 24-hour ambulatory blood pressure monitoring, clinical laboratory safety tests and adverse event assessments will be performed to evaluate the effectiveness of the two doses of vitamin D on blood pressure. Blood samples will be stored for future biomarker assessments. The total duration of the study is anticipated to be 18 months, assuming a 12 month enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 to 50 years of age
* Systolic blood pressure of 120 to 159 mmHg and Diastolic blood pressure ≤99 mmHg
* Vitamin D deficiency, defined as 25-hydroxyvitamin D <25 ng/ml
* No use of any anti-hypertensive medication in last 3 months or anticipated or planned use in next 6 months
* No use of vitamin D supplementation in last 3 months, defined as vitamin D found in a multivitamin or supplement totaling >400 IU per day or anticipated or planned use in next 6 months

Exclusion Criteria:

* Use of any anti-hypertensive medication in last 3 months or anticipated or planned use in next 6 months
* Use of vitamin D supplementation in last 3 months, defined as vitamin D found in a multivitamin or supplement totaling >400 IU per day or anticipated or planned use in next 6 months
* Use of St. John's wart, rifampin, any treatment for HIV, orlistat, oral glucocorticoids, phenobarbital, phenytoin, mineral oil, or bile acid sequestrants in the last 3 months or anticipated or planned use in next 6 months
* Female who is pregnant, nursing, or of childbearing potential and planning or anticipating pregnancy in next 6 months
* History of diabetes mellitus (including Type 1, Type 2 and diet controlled)
* Serum creatinine >2.0 mg/dl or estimated Glomerular Filtration Rate (GFR) <30 ml/min
* Calcium >10.0 mg/dl or phosphorus >5 mg/dl
* History of kidney stones
* Body mass index >38 kg/m2
* Known cardiovascular disease: defined as prior myocardial infarction, percutaneous transluminal coronary angioplasty, coronary artery bypass or stroke
* History of cirrhosis or severe liver disease (defined as history of GI bleeding from liver disease, jaundice or ascites)
* Current heavy alcohol use: defined as drinking 5 or more drinks per occasion on 5 or more days in the past 30 days
* History of ulcerative colitis, Crohn's disease, celiac disease, colostomy, pancreatic enzyme deficiency, short bowel syndrome, gastric bypass, cystic fibrosis, or dumping syndrome.
* Allergy to coconut
* Regular use or planned use of artificial tanning lights in next 6 months
* Use of any investigational product or device in last 3 months or planned use in next 6 months
* Any condition which could limit the ability to complete and comply with 6-month follow up
* Unwillingness or inability to comply with study requirements
* Inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 534 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as the change in mean 24-hour ambulatory systolic blood pressure. | 24 hours

SECONDARY OUTCOMES:
Change in mean 24-hour ambulatory diastolic blood pressure | 24 hours
Change in mean daytime and nighttime ambulatory systolic and diastolic blood pressure | 24 hours
Change in mean clinic systolic and diastolic blood pressure | 6 months
Change in mean clinic pulse pressure | 6 months
Relation of vitamin D status to changes in clinic and 24-hour ambulatory blood pressure measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wang, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota

REFERENCES:
- [Derived] Miao J, Bachmann KN, Huang S, Su YR, Dusek J, Newton-Cheh C, Arora P, Wang TJ. Effects of Vitamin D Supplementation on Cardiovascular and Glycemic Biomarkers. J Am Heart Assoc. 2021 May 18;10(10):e017727. doi: 10.1161/JAHA.120.017727. Epub 2021 May 7. PMID 33960201
- [Derived] Zaleski A, Panza G, Swales H, Arora P, Newton-Cheh C, Wang T, Thompson PD, Taylor B. High-Dose versus Low-Dose Vitamin D Supplementation and Arterial Stiffness among Individuals with Prehypertension and Vitamin D Deficiency. Dis Markers. 2015;2015:918968. doi: 10.1155/2015/918968. Epub 2015 Sep 16. PMID 26451070
- [Derived] Arora P, Song Y, Dusek J, Plotnikoff G, Sabatine MS, Cheng S, Valcour A, Swales H, Taylor B, Carney E, Guanaga D, Young JR, Karol C, Torre M, Azzahir A, Strachan SM, O'Neill DC, Wolf M, Harrell F, Newton-Cheh C, Wang TJ. Vitamin D therapy in individuals with prehypertension or hypertension: the DAYLIGHT trial. Circulation. 2015 Jan 20;131(3):254-62. doi: 10.1161/CIRCULATIONAHA.114.011732. Epub 2014 Oct 30. PMID 25359163